CLINICAL TRIAL: NCT05313178
Title: Acute Changes in Plasma Amino Acid Appearance After Adding Bacillus Coagulans GBI-30, 6086 to Milk Protein Concentrate in Older Women
Brief Title: Changes in Plasma Amino Acid Appearance After Adding Bacillus Coagulans GBI-30, 6086 to Milk Protein Concentrate
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Increnovo, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-21-57
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Protein Malabsorption

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, crossover study design
Who Masked: Participant, Investigator
Masking Description: Supplements blinded to participant and investigator by third party
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milk Protein (Placebo Comparator): 25-gram dose of milk protein concentrate
  Interventions: Dietary Supplement: Bacillus Coagulans GBI-30, 6086
- Milk Protein and Probiotic (Experimental): 25-gram dose of milk protein concentrate with bacillus coagulans GBI-30, 6086
  Interventions: Dietary Supplement: Bacillus Coagulans GBI-30, 6086

INTERVENTIONS:
Dietary Supplement: Bacillus Coagulans GBI-30, 6086 — In a randomized, double-blind, crossover fashion, study participants will supplement on a daily basis for two weeks during one study period with a 25-gram dose of either milk protein concentrate or a 25-gram dose of milk protein concentrate with bacillus coagulans GBI-30, 6086. Each dose will be ingested at the same time of day with 8 - 12 fluid ounces of cold tap water. All participants will be required to complete a supplementation log to document when each dose of their assigned protein is consumed. Upon completion of their first assigned study protocol period, participants will observe a three-week washout period by returning to their normal dietary intake and physical activity habits before beginning supplementation for the remaining study period.

SUMMARY:
The purpose of this study is to examine the pattern of plasma amino acid appearance after a two-week daily regimen of milk protein concentrate supplementation with and without the addition of Bacillus coagulans GBI-30, 6086 among older women.

DETAILED DESCRIPTION:
Once determined eligible and providing consent, participants will be assigned in a randomized, double-blind, crossover fashion to ingest a single daily 25-gram dose of a milk protein concentrate or a similar dose of milk protein concentrate plus bacillus coagulans GBI-30, 6086. Upon arrival for each study visit, participants will have their resting heart rate, blood pressure, body mass, height, and body composition measured. Upon ingestion of their final assigned supplementation dose, standard multiple sample phlebotomy approaches will be used to collect approximately 10mL of venous blood from a forearm vein at specific time intervals up to four hours after ingestion of their final assigned supplementation dose for that period in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between the ages of 50-70 years
* Completing at least 30 minutes of physical activity at minimum three days per week

Exclusion Criteria:

* As indicated on a medical history form they complete, any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, obesity (defined as body mass index > 30 kg/m2), immune, autoimmune, psychiatric, hematological, neurological or endocrinological disorder or disease
* Any woman who is taking a medication known to impact digestive function or hormonal functions that may impact how our body digests, absorbs, or metabolizes nutrients
* Any woman currently taking a probiotic or a dietary supplement that may impact digestive function or hormonal functions that may impact how our body digests, absorbs, or metabolizes nutrients
* Participants who are determined to not be weight stable defined as measured body mass deviating by 2% or more.
* Participants who do not or are not willing to abstain from alcohol, nicotine, and caffeine for overnight (8-10 hours)
* Participants who do not or are not willing to abstain from exercise for 24 hours prior to each visit
* Women who are pregnant
* Women who are lactose intolerant

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of Amino Acids in Blood | 4 hours
  Plasma Concentrations of Amino Acids in Blood

SECONDARY OUTCOMES:
Adverse Events | 4 hours
  Incidence and associations of reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walden KE, Hagele AM, Orr LS, Gross KN, Krieger JM, Jager R, Kerksick CM. Probiotic BC30 Improves Amino Acid Absorption from Plant Protein Concentrate in Older Women. Probiotics Antimicrob Proteins. 2024 Feb;16(1):125-137. doi: 10.1007/s12602-022-10028-4. Epub 2022 Dec 14. PMID 36515888